CLINICAL TRIAL: NCT04987229
Title: Long-term, Safety Extension Study of OLZ/SAM in Pediatric Subjects With Schizophrenia or Bipolar I Disorder
Brief Title: Long-term Safety Extension Study of OLZ/SAM in Pediatric Subjects
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALKS 3831-A313
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Bipolar I Disorder; Schizophrenia
Keywords: Bipolar I Disorder; Schizophrenia; Samidorphan; Pediatric; Olzanzapine; Safety; LYBALVI
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All subjects (Experimental): All subjects will receive OLZ/SAM at a dose determined by the Investigator and based on the olanzapine dosing received in the antecedent study (ALKS 3831-A311 or ALKS 3831-A312 ENLIGHTEN-Youth)
  Interventions: Drug: OLZ/SAM

INTERVENTIONS:
Drug: OLZ/SAM — Olanzapine and Samidorphan fixed dose coated tablet taken once daily
  Other Names: ALKS 3831

SUMMARY:
To evaluate the long-term safety and tolerability of OLZ/SAM in pediatric subjects with schizophrenia or Bipolar I disorder

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed the treatment period in either the ALKS 3831-A311 or the ALKS 3831-A312 study within 10 days of enrolling into this extension study, or subject had terminated early from Study ALKS 3831-A312 due to the clinically significant weight gain criterion.
* Subject will benefit from continued therapy with OLZ/SAM per clinical judgment.
* Subject is able to be treated on an outpatient basis.
* Subject must not be a danger to self or others (per Investigator judgement) and has family support available to be maintained as an outpatient.
* Subject's parent(s)/legal guardian(s) is considered reliable by the Investigator and has agreed to provide support to the subject to ensure compliance with study treatment, visits, and protocol procedures.
* Subject agrees to abide by the contraception requirements specified in the protocol for the duration of the study.

Exclusion Criteria:

* Subject poses a current suicide risk as assessed by the Investigator or as confirmed by the baseline Columbia-Suicide Severity Rating Scale by a response of "Yes" to question numbers 4 or 5 with ideation or suicidal behavior since the last visit.
* Subject has any finding that in the view of the Investigator or Medical Monitor would compromise the safety of the subject or affect their ability to fulfill the protocol visit schedule or visit requirement.
* Subject is currently taking medications that are contraindicated with olanzapine use or exhibit drug-interaction potential with olanzapine
* Subject has a positive test for opioids.
* Subject has a positive urine pregnancy test, is currently pregnant or breastfeeding, or plans to become pregnant or begin breastfeeding at any point during the study and for 90 days after any study drug administration.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 236 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David McDonnell, MD, Study Director — Alkermes, Inc.
Locations (38):
- United States (19):
  - Alkermes Investigational Site, Dothan, Alabama
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Stanford, California
  - Alkermes Investigator Site, Denver, Colorado
  - Alkermes Investigational Site, Washington D.C., District of Columbia
  - Alkermes Investigational Site, Miami, Florida
  - Alkermes Investigational Site, Miami Lakes, Florida
  - Alkermes Investigational Site, Decatur, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Indianapolis, Indiana
  - Alkermes Investigational Site, Saint Charles, Missouri
  - Alkermes Investigational Site, Lincoln, Nebraska
  - Alkermes Investigational Site, Omaha, Nebraska
  - Alkermes Investigational Site, Cincinnati, Ohio
  - Alkermes Investigational Site, West Chester, Ohio
  - Alkermes Investigational Site, DeSoto, Texas
  - Alkermes Investigational Site, Fort Worth, Texas
  - Alkermes Investigational Site, Richmond, Virginia
  - Alkermes Investigational Site, Everett, Washington
- Argentina (5):
  - Alkermes Investigational Site, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Alkermes Investigational Site, La Plata, Buenos Aires
  - Alkermes Investigational Site, Buenos Aires, Buenos Aires F.D.
  - Alkermes Investigational Site, Mendoza, Mendoza Province
  - Alkermes Investigational Site, Córdoba
- Brazil (6):
  - Alkermes Investigational Site, Fortaleza, Ceará
  - Alkermes Investigational Site, Curitiba, Paraná
  - Alkermes Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Alkermes Investigational Site, São Paulo, São Paulo
  - Alkermes Investigational Site, Goiânia
  - Alkermes Investigational Site, São Paulo
- Colombia (4):
  - Alkermes Investigational Site, Barranquilla
  - Alkermes Investigational Site, Bello
  - Alkermes Investigational Site, Bogotá
  - Alkermes Investigational Site, Pereira
- Mexico (4):
  - Alkermes Investigational Site, León, Guanajuato
  - Alkermes Investigational Site, Monterrey, Nuevo León
  - Alkermes Investigational Site, Culiacán, Sinaloa
  - Alkermes Investigational Site, Gustavo A. Madero, State of Mexico

IPD SHARING:
Plan to Share IPD: Undecided